CLINICAL TRIAL: NCT00387881
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Tolerability of TREXIMA* (Sumatriptan Succinate/Naproxen Sodium) for a Single Moderate or Severe Headache in Adults Diagnosed With Probable Migraine Without Aura (ICHD-II 1.6.1) (*TREXIMET)
Brief Title: TREXIMET (Formerly Known as TREXIMA) for the Acute Treatment of Probable Migraine (ICHD-II 1.6.1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TXA107563
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Results first posted 2009-07-10 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Migraine, Without Aura
Keywords: sumatriptan succinate,; naproxen sodium,; parallel group,; double-blind,; placebo-controlled,; Combination product,; migrainous headache; Probable migraine, a sub-type of Migraine; probable migraine,
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treximet (Experimental)
  Interventions: Drug: sumatriptan succinate / naproxen sodium

INTERVENTIONS:
Drug: sumatriptan succinate / naproxen sodium — sumatriptan 85mg / naproxen sodium 500mg
  Arms: Treximet
Drug: Placebo — Placebo to match Treximet tablets
  Arms: Placebo

SUMMARY:
This study was designed to determine the efficacy and tolerability of TREXIMET (formerly known as TREXIMA) compared to placebo for the acute treatment of probable migraine, a sub-type of migraine.

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of probably migraine (6 migraine attacks per month)
* Males and women of childbearing potential on a adequate contraception.

Exclusion Criteria:

* Physician diagnosis of migraine; history of triptan or ergot use; history of headache prophylaxis use
* Pregnant and/or nursing mother
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Basilar or Hemiplegic migraine
* History of stroke or transient ischemic attacks (TIA).
* History of epilepsy or treated with anti-epileptics within the past 5 years.
* Impaired hepatic or renal function.
* History of gastrointestinal bleeding or ulceration.
* Allergy or hypersensitivity to Aspirin or any other NSAID.
* Allergy or hypersensitivity to triptans.
* Participated in an investigational drug trial in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (61):
- United States (61):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Diamond Bar, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valley Stream, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Independence, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Richardson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Silberstein S, Lipton RB, Goldstein J, Aurora SK, White J, Ochs-Ross R, Lener SE, McDonald SA. Evaluation of a New Fixed-dose Single Tablet of Sumatriptan Formulated with RT Technology and Naproxen Sodium (SumaRT/Nap) for the Acute Treatment of Probable Migraine without Aura. Headache 2008: presented at the American Headache Society Meeting, Boston, MA.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TXA107563 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Sumatriptan/Naproxen: Sumatriptan 85 mg and Naproxen sodium 500mg = Treximet (formerly known as Trexima)
Period: Overall Study
Arm/Group | Placebo | Sumatriptan/Naproxen
Started | 334 | 345
Completed | 245 | 243
Not Completed | 89 | 102
Not completed — Lost to Follow-up | 23 | 23
Not completed — Protocol Violation | 2 | 12
Not completed — Withdrawal by Subject | 15 | 18
Not completed — Sponsor terminated Study | 0 | 1
Not completed — Not eligible | 6 | 7
Not completed — No opportunity to treat headache | 32 | 34
Not completed — Not otherwise specified | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Baseline Characteristics used the Safety Population. Not the Randomised Population
- Sumatriptan/Naproxen: Sumatriptan 85 mg and Naproxen sodium 500mg = Treximet. Baseline Characteristics used the Safety Population. Not the Randomised Population
- Total: Total of all reporting groups
Arm/Group | Placebo | Sumatriptan/Naproxen | Total
Number analyzed (Participants) | 246 | 254 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.23) | 35.8 (11.47) | 36.2 (11.35)
Gender [Count of Participants; unit: Participants]
  Female | 176 | 195 | 371
  Male | 70 | 59 | 129
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 28 | 30 | 58
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - East Asian Heritage | 6 | 8 | 14
  Asian - Japanese Heritage | 2 | 1 | 3
  Asian - South East Asian Heritage | 8 | 5 | 13
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African Heritage | 1 | 2 | 3
  White - White/Caucasian/European Heritage | 199 | 206 | 405
  Mixed race | 0 | 1 | 1
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain-Free at 2 Hours Post-dose and Sustained Pain-Free From 2-24 Hours Post-dose.
Description: Pain-free was defined as a headache severity of no pain (grade 0) at 2 hours post-treatment in subjects who have not used rescue medication prior to or at the time of the assessment. Sustained pain-free response was defined as pain-free at 2 hours post-treatment through 24 hours post-treatment without rescue medicine.
Time Frame: 2 hours through 24 hours after Treatment
Population: The Intent to Treat (ITT) Population was the primary analysis population for assessing efficacy and included subjects who treated at least 1 headache attack with randomized treatment and provided at least one post dose evaluation.
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Pain-Free (2 hours) | 25 | 64
  Sustained Pain-Free (2-24 hours) | 20 | 54
Statistical Analysis 1: Comparison: Placebo vs Sumatriptan/Naproxen; Pain-Free (2 hours); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Endpoints were co-primary and both needed to have p-value of <0.05 to be considered indicative of efficacy; Percent difference = 18, 95% CI [10 to 25] — Analysis for Migraine Pain-Free at 2 hours Post-Dose
Statistical Analysis 2: Comparison: Placebo vs Sumatriptan/Naproxen; Sustained Pain-Free (2-24 hours); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percent difference = 15, 95% CI [8 to 22] — Analysis for Sustained Pain Free from 2-24 hours Post-dose

2. Secondary Outcome: Freedom From Headache Pain at 0.5, 1, and 4 Hours After Treatment
Description: Pain-Free is defined as post-treatment headache pain severity of none in subjects who have not used rescue medication prior to or at the time of the assessment.
Time Frame: 0.5, 1, and 4 hours after Treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Pain-free at 4 hours | 60 | 105
  Pain-free at 1 hour | 16 | 23
  Pain-free at 0.5 hour | 6 | 5

3. Secondary Outcome: Sustained Headache Relief 2-24 Hours After Treatment
Description: Sustained pain relief was defined as having pain relief (mild or no pain) at 2 hours w/o any moderate or severe pain during 2-24 hour period post-treatment, without rescue medication.
Time Frame: 2-24 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants | 77 | 110

4. Secondary Outcome: Headache Relief at 4, 2, 1 and 0.5 Hours After Treatment
Description: Pain relief was defined as reduction of headache pain from a baseline severity of moderate or severe to none or mild at the given time.
Time Frame: 0.5, 1, 2, and 4 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Headache relief at 4 hours | 108 | 153
  Headache relief at 2 hours | 113 | 124
  Headache relief at 1 hour | 73 | 85
  Headache relief at 0.5 hour | 39 | 41

5. Secondary Outcome: Subjects Who Used Rescue Medication From 0 - 24 Hours After Treatment
Description: Rescue medication defined as additional medication (i.e. sumatriptan/naproxen sodium as open-label rescue or other medication as permitted per protocol), taken by subject for the treatment of headache pain or other symptoms associated with the headache attack.
Time Frame: 0 - 24 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants | 101 | 61

6. Secondary Outcome: Intermediate Sustained Pain Relief: Post-dose at Intervals of 2-4 Hours and 1-2 Hours After Treatment
Description: Intermediate sustained pain relief was defined as achieving headache pain relief (from moderate or severe pain at baseline to mild or no pain) prior to the specified timepoint (1 or 2 hours) and maintaining it to the specified timepoint (2-4 hours). (Intermediate=Intermed.)
Time Frame: 1-2, and 2- 4 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Intermed. Sustained Pain Relief, 2-4 hrs post-dose | 92 | 118
  Intermed. Sustained Pain Relief, 1-2 hrs post-dose | 67 | 84

7. Secondary Outcome: Intermediate Sustained Pain-Free: Post-dose at Intervals of 2-4 Hours and 1-2 Hours
Description: Intermediate sustained pain free was defined as achieving headache pain-free (moderate or severe pain to no pain) prior to the specified timepoint (1 or 2 hours) and maintaining it to the specified timepoint (2-4 hours).(Intermediate=Intermed.)
Time Frame: 1-2 and 2-4 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Intermed. Sustained Pain-free, 2-4 hrs post-dose | 22 | 61
  Intermed. Sustained Pain-free, 1-2 hrs post-dose | 11 | 23

8. Secondary Outcome: Incidence of Headache Associated: Neck Pain, Sinus Pain, Photophobia, Phonophobia, Nausea at Time Intervals of 4 and 2 Hours After Treatment
Description: Neck pain, sinus pain, photophobia, phonophobia and nausea are considered headache-associated symptoms.(Headache-associated=Headache-Assoc.)
Time Frame: 2 and 4 hours after treatment
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 221 | 222
Participants
  Headache-Assoc. Neck Pain at 4 hours | 93 | 63
  Headache-Assoc. Neck Pain at 2 hours | 68 | 59
  Headache-Assoc. Sinus Pain at 4 hours | 88 | 49
  Headache-Assoc. Sinus Pain at 2 hours | 49 | 36
  Headache-Assoc. Photophobia at 4 hours | 87 | 60
  Headache-Assoc. Photophobia at 2 hours | 60 | 46
  Headache-Assoc. Phonophobia at 4 hours | 83 | 59
  Headache-Assoc. Phonophobia at 2 hours | 53 | 54
  Headache-Assoc. Nausea at 4 hours | 82 | 51
  Headache-Assoc. Nausea at 2 hours | 37 | 36

9. Secondary Outcome: Medication Satisfaction: Mean Patient Perception of Migraine (PPMQ-R) Subscale Score
Description: Patient Perception of Migraine Questionnaire-Revised(PPMQ-R) evaluates subject satisfaction with treatment 24 hours post-dose using validated questions. Questions are analyzed on 4 subscale scores (efficacy, functionality, ease-of-use, and tolerability) and total score. Scores range from 0-100, with the higher scores indicating better satisfaction.
Time Frame: 0 - 24 hours after treatment
Population: ITT Population - Actual numbers of subjects who took questionnaire were Placebo 199 and Sumatriptan/Naproxen=188
Measure: Mean (Standard Error); unit: Score in scale
Arm/Group | Placebo | Sumatriptan/Naproxen
Number analyzed (Participants) | 199 | 188
Score in scale
  Efficacy Adjusted Mean | 53 (2.0) | 67 (2.0)
  Functionality Adjusted Mean | 56 (2.1) | 70 (2.1)
  Ease-of-Use Adjusted Mean | 84 (1.3) | 88 (1.3)
  Bothersome-of-Side Effects Adjusted Mean | 94 (0.8) | 91 (0.8)
  Total Score adjusted Mean | 64 (1.5) | 75 (1.6)

ADVERSE EVENTS:
Arm/Group | Placebo | Sumatriptan/Naproxen
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/254
Other Adverse Events (participants affected / at risk) | 0/246 | 0/254

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the Publication of results from all centers of a multi-center trial but requests that reports based on Single-site data not precede the primary publication of the entire clinical trial.